CLINICAL TRIAL: NCT06031402
Title: Timing of Endoscopy in Cirrhotic Patients with Acute Variceal Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHNKKY-ENDO-AVB
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Upper Gastrointestinal Bleeding; Acute Variceal Bleeding
Keywords: liver cirrhosis; variceal bleeding; gastrointestinal bleeding; endoscopy; survival; randomized controlled trial
MeSH Terms: conditions — Liver Cirrhosis; Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Before enrollment, all patients and/or their relatives will be informed about the study protocol, and sign the written informed consent forms. Eligible patients are randomly assigned at a ratio of 1:1 to early endoscopy group (within 12 hours after admission) and delayed endoscopy group (within 12-24 hours after admission)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early endoscopy group (Experimental): Intervention of endoscopy is within 12 hours after admission
  Interventions: Procedure: Endoscopy
- Delayed endoscopy group (Active Comparator): Intervention of endoscopy is within 12-24 hours after admission
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopy

SUMMARY:
Endoscopy is important for the diagnosis and treatment of acute upper gastrointestinal bleeding (AUGIB), especially acute variceal bleeding (AVB), in patients with liver cirrhosis. However, the optimal timing of endoscopy remains controversial, primarily because the currently available evidence is of poor quality, and the definition of early endoscopy is also very heterogeneous among studies. Herein, a multicenter randomized controlled trial (RCT) is performed to explore the impact of timing of endoscopy on the outcomes of cirrhotic patients with AVB.

DETAILED DESCRIPTION:
A total of 368 cirrhotic patients presenting with AUGIB that is highly suspected to be from AVB will be enrolled. They will be stratified according to the severity of liver function and hemodynamic status at admission, and randomly assigned at a 1:1 ratio into early (within 12 hours after admission) and delayed (within 12-24 hours after admission) endoscopy groups within each stratum. The primary outcomes include the rates of 5-day failure to control bleeding after admission and 6-week rebleeding. The secondary outcomes include 6-week mortality and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. patients with AUGIB which is highly suspected to be caused by gastroesophageal variceal rupture;
2. patients with a diagnosis of liver cirrhosis based on imaging and pathology;
3. patients and/or their relatives who sign informed consents;
4. patients' age ≥18 years.

Exclusion Criteria:

1. patients who have undergone endoscopy at other hospitals before admissions;
2. patients' hemodynamics are unstable after resuscitation;
3. patients with severe cardiovascular or cerebrovascular diseases or renal injury;
4. patients who have taken anticoagulants or antiplatelet drugs within 2 weeks before admissions, or are diagnosed with severe hematological diseases;
5. patients with human immunodeficiency virus or other acquired or congenital immune deficiency diseases;
6. patients with mental illness;
7. pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The failure to control bleeding after admissions | within 5 days admission
  Failure to control bleeding is defined as any one of the three following conditions within 5 days admission: 1) vomiting of fresh blood; 2) suction of more than 100ml of fresh blood from the nasogastric tube; 3) a decrease in hemoglobin concentration of 30g/L in the absence of blood transfusion; or 4) death.
6-week rebleeding | 6-week
  Rebleeding is defined as new onset of hematemesis or melena after successful treatment.

SECONDARY OUTCOMES:
6-week all-cause mortality | 6-week
  Death.
Adverse events | up to 6 weeks
  Adverse events include fever, chest pain, dysphagia, and perforation or pneumonia caused by endoscopy or anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, MD, Principal Investigator — General Hospital of Shenyang Military Area; Yiling Li, MD, Principal Investigator — First Hospital of China Medical University; Bimin Li, MD, Principal Investigator — The First Affiliated Hospital of Nanchang University; Xuefeng Luo, MD, Principal Investigator — West China Hospital; Xiaofeng Liu, MD, Principal Investigator — The 960th Hospital of the Chinese People's Liberation Army; Chunqing Zhang, MD, Principal Investigator — Affiliated Provincial Hospital of Shandong First Medical University; Mingkai Chen, MD, Principal Investigator — People's Hospital of Wuhan University; Derun Kong, MD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Fernando G Romeiro, MD, Principal Investigator — Botucatu Medical School; Andrea Mancuso, MD, Principal Investigator — Azienda di Rilievo Nazionale ad Alta Specializzazione Civico-Di Cristina-Benfratelli; Nahum Méndez-Sánchez, MD, Principal Investigator — Medica Sur Clinic and Foundation; Enqiang Linghu, MD, Principal Investigator — The First Medical Center of Chinese PLA General Hospital; Yunhai Wu, MD, Principal Investigator — The Sixth People&amp;#39;s Hospital of Shenyang; Metin Basaranoglu, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Z, Wang R, Cheng G, Ma D, Ibrahim M, Chawla S, Qi X. Outcomes of early versus delayed endoscopy in cirrhotic patients with acute variceal bleeding: a systematic review with meta-analysis. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e868-e876. doi: 10.1097/MEG.0000000000002282. PMID 35048654
- [Background] Peng Y, Qi X, Dai J, Li H, Guo X. Child-Pugh versus MELD score for predicting the in-hospital mortality of acute upper gastrointestinal bleeding in liver cirrhosis. Int J Clin Exp Med. 2015 Jan 15;8(1):751-7. eCollection 2015. PMID 25785053
- [Background] Peng Y, Qi X, Guo X. Child-Pugh Versus MELD Score for the Assessment of Prognosis in Liver Cirrhosis: A Systematic Review and Meta-Analysis of Observational Studies. Medicine (Baltimore). 2016 Feb;95(8):e2877. doi: 10.1097/MD.0000000000002877. PMID 26937922
- [Background] Li Y, Li H, Zhu Q, Tsochatzis E, Wang R, Guo X, Qi X. Effect of acute upper gastrointestinal bleeding manifestations at admission on the in-hospital outcomes of liver cirrhosis: hematemesis versus melena without hematemesis. Eur J Gastroenterol Hepatol. 2019 Nov;31(11):1334-1341. doi: 10.1097/MEG.0000000000001524. PMID 31524777
- [Derived] Qi X, Li Y, Li B, Luo X, Liu X, Zhang C, Chen M, Kong D, Wu Y, Romeiro FG, Basaranoglu M, Zhang J, Li Q, Wang R, Shao X, Guan L, Wang N, You Y, He M, Wang X, Huang J, Wu W, Li Q, Zhang M, Wang G, Zhang C, Cheng D, Zhang Q, Mei X, Sun N, Ban Y, Marcondes MB, Yamashiro FDS, Mutlu E, Zheng Z, Peng M, Xu W, Li Z, Chai L, Linghu E. Timing of endoscopy in cirrhotic patients with acute variceal bleeding: protocol of a multicenter randomized controlled trial. Therap Adv Gastroenterol. 2024 Nov 13;17:17562848241295452. doi: 10.1177/17562848241295452. eCollection 2024. PMID 39539489